CLINICAL TRIAL: NCT01393886
Title: A Prospective, Open-label Study to Evaluate the Safety and Efficacy of Laparoscopic Greater Curvature Plication (LGCP) in the Treatment of Obese Patients
Brief Title: LGCP (Laparoscopic Greater Curvature Plication)
Acronym: LGCP
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Principal Investigator, Heekoung A Youn, Research coordinator, NYU Langone Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R11-00797
Record Dates: First submitted 2011-06-09; First posted 2011-07-13 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Obesity
Keywords: Obesity Surgery
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Laparoscopic Greater Curvature Plication (Experimental): Only one treatment arm
  Interventions: Procedure: Laparoscopic Greater Curvature Plication (LGCP)

INTERVENTIONS:
Procedure: Laparoscopic Greater Curvature Plication (LGCP) — This procedure creates a small sized stomach by folding the stomach twice into itself vertically. The functional capacity of the stomach is decreased by 80% of its normal(At least two rows of five continuous stitches are placed laparoscopically about the greater curvature of the stomach starting at or near the angle of His and ending in the antrum).

SUMMARY:
The aim of this study is to find out the safety and efficacy of Laparoscopic Greater Curvature Plication (LGCP) procedure. This study procedure is an alternative restrictive weight loss surgery that has the potential to reduce the complications associated with gastric banding and sleeve gastrectomy by creating a small sized stomach without the use of an implant and without cutting stomach.

DETAILED DESCRIPTION:
STUDY OBJECTIVES: To demonstrate the safety and efficacy of Laparoscopic Greater Curvature Plication (LGCP)

DESIGN: Prospective, open-label, and single center

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years of age at the time of enrollment into the study;
* Have a BMI of at least 30;
* Subject is willing to give consent and comply with protocol evaluation and treatment schedules;
* Subject agrees to refrain from any type of weight-loss drug (prescription or OCT) or elective procedure that affect body weight for the duration of the trial; and
* HbA1C<11%

Exclusion Criteria:

* History of previous malabsorptive bariatric procedures;
* Women of childbearing potential who are pregnant or lactating at the time of screening or at the time of surgery;
* Any condition which precludes compliance with the study;
* History or presence of pre-existing autoimmune connective tissue disease; and
* Use of prescription or over the counter weight reduction medications or supplements within 30 days of the screening visit or the duration of study participation.

This study is a local study (NY, within 50 miles). This study is not a sponsored trial. Therefore, the procedure is not free.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-06; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Weight Loss | 12 months
  The primary effectiveness endpoint is % of subjects who attain clinically successful weight loss at one year post LGCP.

SECONDARY OUTCOMES:
Morbidity rates | 12 months
  Morbidity rates
Mortality rates | 12 month
  Mortality rates

CONTACTS AND LOCATIONS:
Overall Officials: Fielding George, M.D., Principal Investigator — NYU SOM; Christine Fielding, M.D., Principal Investigator — NYU SOM; Marina Kurian, M.D., Principal Investigator — NYU SOM
Locations (1):
- NYU Langone Medical Center, New York, New York, United States

REFERENCES:
- [Result] Ramos A, Galvao Neto M, Galvao M, Evangelista LF, Campos JM, Ferraz A. Laparoscopic greater curvature plication: initial results of an alternative restrictive bariatric procedure. Obes Surg. 2010 Jul;20(7):913-8. doi: 10.1007/s11695-010-0132-0. PMID 20407932
- See also: Related Info — http://thinforlife.med.nyu.edu/research/clinical-trials